CLINICAL TRIAL: NCT02041507
Title: A Randomized, Controlled Trial Comparing Air Insufflation, Water Immersion and Water Exchange for Adenoma Detection Rate in Screening Colonoscopy
Brief Title: Water-aided Colonoscopy vs Air Insufflation Colonoscopy in Colorectal Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Presidio Ospedaliero Santa Barbara (Other)
Responsible Party: Principal Investigator, Sergio Cadoni, M.D., Responsabile Servizio Endoscopia Digestiva, Presidio Ospedaliero Santa Barbara
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: PI.2013.2502; Delibera 1047.2013 (Other: ASL 07 Carbonia, Italy)
Record Dates: First submitted 2014-01-18; First posted 2014-01-22 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Colorectal Cancer; Colorectal Adenomas; Colorectal Polyps; Pain
Keywords: Water-aided colonoscopy; Water Immersion; Water Exchange; On-demand sedation; Unsedated colonoscopy; Adenoma detection rate; Mean adenomas per procedure
MeSH Terms: conditions — Colorectal Neoplasms; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Air insufflation method. (Active Comparator): Colonoscopy performed in the standard fashion, with the minimal air insufflation required to aid insertion and allowing for washing as needed. Considered to be standard procedure.
  Interventions: Other: Air insufflation method.
- Water Immersion method. (Experimental): Infusion of water during the insertion phase of colonoscopy mainly to open the colonic lumen and progress to the cecum immersed in the water environment thus created, without attempting to clear the colon contents. Residual air in the colon will not be removed. Infused water and residual feces will be suctioned back predominantly during withdrawal. Insufflation not used until the cecum is reached. It will be allowed only 3 times and no more than 10 seconds each time (ITT failure if >3) if the lumen cannot be seen. Withdrawal phase done using air insufflation.
  Interventions: Other: Water Immersion method.
- Water Exchange method. (Experimental): Insufflation not used until the cecum is reached. Infusion of a sufficient amount of water to render the lumen of the colon a slit to progress with the colonoscope. Part of the infused water will be constantly suctioned back exchanging clean for dirty or hazy water. Air pockets will be always aspirated to collapse the lumen. After cecal intubation as much residual water as possible will be aspirated before beginning the withdrawal phase. During withdrawal residual water and feces will be suctioned. Withdrawal phase done using air insufflation.
  Interventions: Other: Water Exchange method.

INTERVENTIONS:
Other: Air insufflation method. — Air insufflation colonoscopy.
  Arms: Air insufflation method.
Other: Water Immersion method. — Water Immersion during insertion, air insufflation during withdrawal.
  Arms: Water Immersion method.
Other: Water Exchange method. — Water Exchange during insertion, air insufflation during withdrawal.
  Arms: Water Exchange method.

SUMMARY:
The degree of protection afforded by colonoscopy against proximal colorectal cancer (CRC) appears to be related to the quality of the procedure, and the incomplete removal of lesions has been shown to increase the subsequent risk of developing a colon cancer.

Some studies suggest that small polyps with advanced histology are more common in the right than in the left colon (right colon proximal to splenic flexure, left colon distal to the splenic flexure). The average size of polyps in the right colon with advanced pathology or containing adenocarcinoma was ≤9 mm, whereas in the left colon their average size was >9 mm, P<0.001. Inadequate prevention of right-sided CRC incidence and mortality may be due to right-sided polyps with advanced histology or that harbor malignancy. These presumptive precursors of cancer are smaller and possibly more easily obscured by residual feces, and more likely to be missed at colonoscopy.

Water-aided colonoscopy (WAC) can be subdivided broadly into two major categories: water immersion (WI), characterized by suction removal of the infused water predominantly during the withdrawal phase of colonoscopy, and water exchange (WE), characterized by suction removal of infused water predominantly during the insertion phase of colonoscopy.

In some reports WE appeared to be superior to both WI and air insufflation colonoscopy (AI) in terms of pain reduction and adenoma detection, particularly for <10 mm adenomas in the proximal colon.

In this multicenter, double-blinded randomized controlled trial (RCT) we test the hypothesis that that WE, compared to AI and WI, will enhance overall Adenoma Detection Rate (ADR) in CRC screening patients. Confirmation of the primary hypothesis will provide evidence that WE enhances the quality of screening colonoscopy.

We also hypothesize that WE may be more effective in detecting proximal colon adenomas than WI and AI, particularly <10 mm adenomas, thus increasing proximal colon ADR and proximal colon ADR <10 mm. Confirmation of secondary hypotheses will provide justification for further testing that WE may provide a strategy to improve prevention of colorectal cancer by increasing detection of adenomas in screening colonoscopy.

Unlike previous reports of single colonoscopist studies, the insertion and withdrawal phases of colonoscopy will be done by different investigators. The second investigator will be blinded to the method used to insert the instrument, thus eliminating possible bias about procedure related issues.

Several secondary outcomes will also be analysed.

DETAILED DESCRIPTION:
Design: Prospective double-blinded multicenter randomized controlled trial. Methods: Colonoscopy with Air Insufflation, Water Immersion, Water Exchange to aid insertion of colonoscope; split dose bowel preparation. Sedation available at the start of the procedure or on-demand.

Control method: Air insufflation colonoscopy. Study methods: Water Immersion colonoscopy, Water Exchange colonoscopy.

Population: Consecutive 50 to 70 year-old screening patients. After informed consent, assignment to control or study arms based on computer generated randomization list with block allocation and stratification.

Primary outcome: overall Adenoma Detection Rate. Secondary outcomes: proximal colon ADR, Mean Adenomas resected per Procedure (MAP), cecal intubation rate and time, total procedure time (including biopsy and/or polypectomy), maximum pain during colonoscopy assessed during insertion and at discharge, the need for sedation/analgesia and its dosage. In addition loop reduction maneuvers, position changes, abdominal compression, the amount of infused and suctioned water during insertion and withdrawal, and patients willingness to repeat the examination will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* consecutive screening patients

Exclusion Criteria:

* previous colonoscopy within 5 years
* surveillance colonoscopy
* previous colorectal surgery
* indication for a proctosigmoidoscopy or bidirectional endoscopy
* history of inflammatory bowel disease
* patient refusal or inability to provide informed consent
* inadequate consumption of bowel preparation

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1224 (Actual)
Dates: Start 2014-02; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Adenoma Detection Rate. | 18 months.
  Proportion of subjects with at least one adenoma of any size.

SECONDARY OUTCOMES:
Proximal colon Adenoma Detection Rate. | 18 months.
  Proportion of subjects with at least one adenoma of any size in the proximal colon.
Proximal colon <10 mm Adenoma Detection Rate. | 18 months.
  Proportion of subjects with at least one adenoma <10 mm in the proximal colon.
Mean adenomas resected per procedure. | 18 months.
  Total number of adenomas resected per subject.
Cecal intubation rate. | 1 hour.
  Cecal intubation will be defined as passage of the tip of the colonoscope beyond the ileocecal valve so that the medial wall of the cecum proximal to the ileocecal valve will be observed.
Cecal intubation time. | 1 hour.
  Cecal intubation time will be defined as the time for passage of the colonoscope from the rectum to the cecum.
Total procedure time. | 1 hour.
  Total procedure time (including time required for polyp resection or biopsy).
Maximum pain score recorded during insertion phase of colonoscopy. | 1 hour.
  Pain will be measured on a visual analogue scale (VAS) with a score 0=absence of pain, 1-2=simply "discomfort", 10=the worst possible pain. Before the procedure, an endoscopic nurse will explain the VAS scoring system to the patient. Patient will be informed that the request for pain information is not to remind that the examination should be uncomfortable, but to let the colonoscopist be alerted to the need to use maneuvers to minimize discomfort (e.g. loop reduction, removal of colonic content, abdominal compression and/or change in patient position). At regular intervals during colonoscopy (e.g. every 60 seconds) patients will be asked about discomfort or pain. The responses will be recorded, and the maximum pain score noted.
Pain score at discharge. | 1 hour.
  After the procedure and at discharge from the Endoscopy Unit, an assistant nurse blinded to the procedure will ask patients about maximum pain during insertion phase of the procedure using the same VAS when neither the endoscopist nor the assistant nurse who performed the colonoscopy will be present. Patients will be asked to quantify the degree of pain experienced and to place a mark over the VAS accordingly.
Need for sedation/analgesia and its dosage | 1 hour.
  All patients will be offered sedation for the procedure. Patients can accept or decline the medication. If they accept, the procedure will be started with the administration of 2 mg of Midazolam intravenously (minimal sedation). If the patient will choose on-demand sedation, minimal sedation will be offered when pain score reaches ≥2 on the VAS. Patients can accept or decline the offered medication. If they accept, minimal sedation will be administered as described above. To avoid bias by the colonoscopist, sedation medication will be administered based on the patients' confirmation that the pain is no longer tolerable, and not at the discretion of the colonoscopist. The colon segment in which patients requests sedation will be recorded. If additional medication will be required despite the abovementioned maneuvers and/or minimal sedation, it will be provided according to local standards and it will be recorded.

OTHER OUTCOMES:
Loop reduction maneuvers. | 1 hour.
  Applied as needed if advancement of the colonoscope fails.
Position changes. Position changes. Position changes. Position changes. Position changes. | 1 hour.
  Change in patient position as needed if advancement of the colonoscope fails.
Abdominal compression. | 1 hour.
  Compression of abdomen if advancement of the colonoscope fails.
Amount of water used during the procedure. | 1 hour.
  Amount of water infused and aspirated during insertion and withdrawal.
Patients willingness to repeat the examination. | 1 hour.
  Patients willingness to repeat the examination based on overall satisfaction about procedure. Measured at discharge on a yes/no question.

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Cadoni, MD, Principal Investigator — S. Barbara Hospital, Iglesias (CI), Italy
Locations (4):
- Sepulveda Ambulatory Care Center, VA Greater Los Angeles Healthcare System, Los Angeles, California, United States
- Digestive Diseases Center, Vìtkovice Hospital, Ostrava, Czechia
- Italy (2):
  - Digestive Endoscopy Unit, Ospedale S. Barbara, Iglesias, CI
  - Division of Gastroenterology, Ospedale Valduce, Como, CO

REFERENCES:
- [Background] Leung FW, Amato A, Ell C, Friedland S, Harker JO, Hsieh YH, Leung JW, Mann SK, Paggi S, Pohl J, Radaelli F, Ramirez FC, Siao-Salera R, Terruzzi V. Water-aided colonoscopy: a systematic review. Gastrointest Endosc. 2012 Sep;76(3):657-66. doi: 10.1016/j.gie.2012.04.467. PMID 22898423
- [Background] Gupta S, Balasubramanian BA, Fu T, Genta RM, Rockey DC, Lash R. Polyps with advanced neoplasia are smaller in the right than in the left colon: implications for colorectal cancer screening. Clin Gastroenterol Hepatol. 2012 Dec;10(12):1395-1401.e2. doi: 10.1016/j.cgh.2012.07.004. Epub 2012 Jul 24. PMID 22835574
- [Background] Cadoni S, Gallittu P, Sanna S, Fanari V, Porcedda ML, Erriu M, Leung FW. A two-center randomized controlled trial of water-aided colonoscopy versus air insufflation colonoscopy. Endoscopy. 2014 Mar;46(3):212-8. doi: 10.1055/s-0033-1353604. Epub 2013 Nov 11. PMID 24218307
- [Background] Radaelli F, Paggi S, Amato A, Terruzzi V. Warm water infusion versus air insufflation for unsedated colonoscopy: a randomized, controlled trial. Gastrointest Endosc. 2010 Oct;72(4):701-9. doi: 10.1016/j.gie.2010.06.025. PMID 20883846
- [Background] Leung FW. Water-aided colonoscopy. Gastroenterol Clin North Am. 2013 Sep;42(3):507-19. doi: 10.1016/j.gtc.2013.05.006. PMID 23931857
- [Background] Rabenstein T, Radaelli F, Zolk O. Warm water infusion colonoscopy: a review and meta-analysis. Endoscopy. 2012 Oct;44(10):940-51. doi: 10.1055/s-0032-1310157. Epub 2012 Sep 17. PMID 22987214
- [Derived] Cadoni S, Falt P, Rondonotti E, Radaelli F, Fojtik P, Gallittu P, Liggi M, Amato A, Paggi S, Smajstrla V, Urban O, Erriu M, Koo M, Leung FW. Water exchange for screening colonoscopy increases adenoma detection rate: a multicenter, double-blinded, randomized controlled trial. Endoscopy. 2017 May;49(5):456-467. doi: 10.1055/s-0043-101229. Epub 2017 Mar 10. PMID 28282689